CLINICAL TRIAL: NCT00000581
Title: Granulocyte Transfusion Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: 301; N01-HB-6-2970 (Other Grant/Funding Number: US NIH Contract Number); N01-HB-6-2971 (Other Grant/Funding Number: US NIH Contract Number); N01-HB-6-2972 (Other Grant/Funding Number: US NIH Contract Number); N01-HB-6-2973 (Other Grant/Funding Number: US NIH Contract Number)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2000-01

CONDITIONS: Blood Transfusion; Infection
MeSH Terms: conditions — Infections | interventions — Leukocyte Transfusion

INTERVENTIONS:
Procedure: leukocyte transfusions

SUMMARY:
To evaluate granulocyte transfusion therapy with respect to its prophylactic and therapeutic effectiveness to prevent and aid recovery from infection. The study trials were conducted simultaneously.

DETAILED DESCRIPTION:
BACKGROUND:

Infection remains a major cause of death in patients receiving chemotherapy for malignant diseases. One approach to the problem of septicemia and high mortality in these patients was the therapeutic use of granulocyte transfusions. Improvements in collection techniques, employing continuous flow centrifugation, permitted the collection of granulocytes from a single, normal donor in sufficient numbers to study their application in the treatment of infections in granulocytopenic patients. Studies had demonstrated the efficacy of granulocyte transfusions as an adjunct in the therapy of septicemia due to gram negative microorganisms associated with granulocytopenia.

The aims of the study were to determine (1) whether infections could be prevented in patients who received granulocytes prophylactically and (2) whether recovery from infection was aided in patients who received granulocytes therapeutically. Both trials utilized controls who received no granulocytes.

Four contracts were awarded in September 1976. The protocol designed to evaluate the efficacy of prophylactic granulocyte transfusions was completed at the close of 1977. The protocol for the therapeutic trial was completed in April 1978. Approximately 90 patients were randomized in the prophylactic trial and 51 in the therapeutic trial. The Recruitment and Intervention Phase ended in February 1980. The trial has concluded.

DESIGN NARRATIVE:

Prophylactic Trial and Therapeutic Trial: randomized, non-blind, sequential. Eligible patients were randomized to daily granulocyte transfusions or no granulocyte transfusions.

The study completion date listed in this record was inferred from the first publication listed in the Citations section of this study record.

ELIGIBILITY:
Prophylactic Trial: males and females, 12 years or older, who were in the first induction phase of chemotherapy for acute leukemia, who had severe neutropenia, and who did not have documented infection.

Therapeutic Trial: males and females, any

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1976-09; Study Completion 1981-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Gale — University of California; Geoffrey Herzig — Washington University School of Medicine; Ronald Strauss — University of Iowa

REFERENCES:
- [Background] Strauss RG, Connett JE, Gale RP, Bloomfield CD, Herzig GP, McCullough J, Maguire LC, Winston DJ, Ho W, Stump DC, Miller WV, Koepke JA. A controlled trial of prophylactic granulocyte transfusions during initial induction chemotherapy for acute myelogenous leukemia. N Engl J Med. 1981 Sep 10;305(11):597-603. doi: 10.1056/NEJM198109103051101. PMID 6790985
- [Background] Winston DJ, Ho WG, Gale RP. Prophylactic granulocyte transfusions during chemotherapy of acute nonlymphocytic leukemia. Ann Intern Med. 1981 May;94(5):616-22. doi: 10.7326/0003-4819-94-5-616. PMID 6263139